CLINICAL TRIAL: NCT06839534
Title: The Effects of Maternal Voice Listening Program on Preterm Infant Responses and Maternal-Infant Attachment in the Neonatal Intensive Care Unit
Brief Title: Effects of a Structured Maternal Voice Program on Premature Infant Responses and Maternal-Infant Attachment in the Neonatal Intensive Care Unit
Acronym: SMVP-NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Queen Sirikit National Institute of Child Health (QSNICH), Thailand (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: REC.097/2024
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Neonatal Intensive Care Unit; PreTerm Neonate; Healthy
Keywords: Premature Infants; Neonatal Intensive Care Unit; Maternal-Infant Attachment; Infant Behavioral Responses; Maternal Voice
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: This study uses a quasi-experimental crossover design to evaluate the effects of the Structured Maternal Voice Program (SMVP) on premature infant responses and maternal-infant attachment. Participants are randomly assigned to two sequences: (1) SMVP intervention followed by standard nursing care, or (2) standard nursing care followed by SMVP intervention. A one-day washout period is included between crossover phases to minimize residual effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Maternal Voice Program (SMVP) (Experimental): Participants in this group receive the Structured Maternal Voice Program (SMVP) for four days, followed by standard nursing care for four days after a one-day washout period.
  Interventions: Behavioral: Structured Maternal Voice Program (SMVP)
- Standard Nursing Care (Other): Participants in this group receive standard nursing care for four days, followed by the Structured Maternal Voice Program (SMVP) for four days after a one-day washout period.
  Interventions: Behavioral: Structured Maternal Voice Program (SMVP)

INTERVENTIONS:
Behavioral: Structured Maternal Voice Program (SMVP) — Pre-recorded maternal voice messages played via an MP3 player integrated into the infant's incubator. The recordings include recognition messages ("I'm so glad to have you") and soothing messages ("Rest well, little one, you're safe with me"). The intervention is delivered three times daily for five minutes per session over a four-day period.

SUMMARY:
This study evaluates the effects of a Structured Maternal Voice Program (SMVP). on premature infant responses and maternal-infant attachment in the intensive care unit (NICU) . Using a quasi-experimental crossover design, 16 mother-infant pairs (gestational age 32-36 weeks) were randomly assigned to experimental or control phases, with a four-day intervention and a one-day washout period. Infant responses and attachment outcomes were assessed using validated tools. Findings indicate significant improvements in motor activity, sleep states, and maternal-infant attachment scores, supporting the integration of maternal voice interventions in neonatal care.

DETAILED DESCRIPTION:
Background & Rationale Premature infants in the Neonatal Intensive Care Unit (NICU) face significant developmental challenges due to maternal separation and environmental stressors, such as excessive noise, bright lights, and invasive medical procedures. These stressors can negatively affect biobehavioral responses, including sleep-wake patterns, motor activity, and physiological stability. Moreover, the absence of maternal presence in NICUs can impair the maternal-infant attachment process, which is crucial for emotional bonding and neurodevelopment.

The Structured Maternal Voice Program (SMVP) is an innovative intervention designed to address these challenges by exposing preterm infants to their mother's voice through pre-recorded audio messages. This program is based on existing evidence that supports the role of maternal voice in stabilizing neonatal responses, promoting sleep regulation, and enhancing attachment. However, limited research has been conducted on the structured implementation of maternal voice exposure in NICUs, especially in settings where maternal visitation is restricted.

This study aims to evaluate the effectiveness of the SMVP in improving premature infant biobehavioral responses and maternal-infant attachment in a NICU setting.

Study Objectives

The primary objectives of this study are to:

Evaluate the impact of SMVP on premature infant responses, including motor activity, behavioral states, and sleep-wake patterns.

Assess changes in maternal-infant attachment scores before and after exposure to SMVP.

Study Design This study is a quasi-experimental crossover trial conducted at the Queen Sirikit National Institute of Child Health (QSNICH), Bangkok, Thailand. The study is designed to minimize confounding variables using a crossover design involving two groups.

Participants: 16 mother-infant pairs (infants born at 32-36 weeks gestational age) Randomization: Infants are randomly assigned to either the experimental phase (SMVP first) or the control phase (standard nursing care first) Washout Period: A one-day washout period between crossover sequences to prevent residual effects from the initial phase Duration: The intervention lasts four consecutive days per phase Intervention Details

The Structured Maternal Voice Program (SMVP) involves playing pre-recorded maternal voice messages through an MP3 player integrated into the incubator. The voice recordings consist of:

Recognition messages: Short affirmations such as "I'm so glad to have you." Soothing messages: Longer comforting phrases such as "Rest well, little one, you're safe with me."

Playback schedule:

Three times daily (morning, afternoon, and evening) Five-minute duration per session Calibrated at 55-60 dB to mimic intrauterine auditory experiences The control group receives standard nursing care without maternal voice exposure during the initial phase. After the washout period, the groups switch interventions.

Outcome Measures

Primary Outcomes:

Infant motor activity: including single limb movement, gross body movement, and head movement Infant behavioral states: including active sleep and quiet alert

Secondary Outcome:

Maternal-Infant Attachment Score, measured using the Maternal-Infant Attachment Questionnaire Significance

The findings from this study may:

Provide empirical evidence supporting the use of maternal voice exposure in NICUs as a structured intervention.

Offer a non-invasive, cost-effective intervention that enhances preterm infant stability and development.

Contribute to the integration of maternal voice programs into routine NICU care to improve outcomes for preterm infants.

Serve as a model for addressing maternal-infant separation in settings with restricted hospital visitation, ensuring both emotional and developmental needs are met for preterm infants.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants born at 32-36 weeks gestational age
2. Receiving care in the Neonatal Intensive Care Unit (NICU) at QSNICH
3. Stable vital signs with no severe medical complications that would interfere with auditory perception
4. Mothers willing and able to provide pre-recorded voice messages for SMVP
5. Parental informed consent obtained

Exclusion Criteria:

1. Critically unstable infants with severe medical complications (e.g., respiratory failure, severe metabolic acidosis)
2. Infants with diagnosed auditory or neurological impairments affecting response to maternal voice
3. Infants with severe intraventricular hemorrhage (Grade III or higher)
4. Mothers unable to provide pre-recorded voice messages due to health or psychological limitations
5. Families declining participation or withdrawing consent

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Premature Infant Responses | Four days of intervention per phase
  Premature infant responses, including motor activity and behavioral states, will be assessed before, during, and after exposure to the Structured Maternal Voice Program (SMVP). The assessment will include:
  * Motor Activity: Single limb movement, gross body movement, head movement
  * Behavioral States: Active sleep, quiet alert Observations will be conducted by trained NICU nurses using a standardized Infant Response Assessment Tool. Responses will be recorded during each intervention phase and analyzed using repeated measures analysis.

SECONDARY OUTCOMES:
Maternal-Infant Attachment Score | Before and after the intervention phase (4 days per phase)
  Maternal-infant attachment will be assessed before and after exposure to the Structured Maternal Voice Program (SMVP) using the Maternal-Infant Attachment Questionnaire (MIAQ). This validated tool measures maternal bonding and emotional connection with the infant, evaluating factors such as maternal sensitivity, affectionate behaviors, and perceived closeness. The questionnaire will be administered to mothers on Day 1 (pre-intervention) and Day 4 (post-intervention) of each phase. Statistical analyses will compare changes in attachment scores across conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Surasak Treenai Faculty of Nursing, Chulalongkorn University, Ph.D., Nursing, Principal Investigator — Faculty of Nursing, Chulalongkorn University
Locations (1):
- Faculty of Nursing, Chulalongkorn University, Bangkok, Patumwan, Thailand

IPD SHARING:
Plan to Share IPD: No
Due to ethical considerations and the sensitive nature of neonatal and maternal-infant attachment data, individual participant data (IPD) will not be shared publicly. However, aggregated and de-identified results will be published in peer-reviewed journals and presented at scientific conferences.

REFERENCES:
- [Background] Filippa M, Panza C, Ferrari F, Frassoldati R, Kuhn P, Balduzzi S, D'Amico R. Systematic review of maternal voice interventions demonstrates increased stability in preterm infants. Acta Paediatr. 2017 Aug;106(8):1220-1229. doi: 10.1111/apa.13832. Epub 2017 Apr 19. PMID 28378337
- See also: Institutional Review Board (IRB) of Queen Sirikit National Institute of Child Health (QSNICH): Ethical approval and research guidelines. — https://sites.google.com/view/researchqsnich/%E0%B8%AB%E0%B8%99%E0%B8%B2%E0%B9%81%E0%B8%A3%E0%B8%81?authuser=4